CLINICAL TRIAL: NCT06462638
Title: Study on the Developmental Value of the Physical and Vocal Contact Relationship Between Preterm Infant in the NICU and Caregivers (Mother, Father, Nurse)
Brief Title: COntact RElationship in Neonatal Intensive Care Unit
Acronym: CORE in NICU
Status: Recruiting | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Scienze Psicologiche,Pedagogiche,Università degli Studi di Palermo (Unknown); UOC Neonatologia e UTIN, Presidio Ospedaliero G. F. Ingrassia di Palermo (Unknown)
Responsible Party: Principal Investigator, Gennaro Tartarisco, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2024-007
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth; Postpartum Depression
Keywords: preterm birth; contact relationship; postpartum depression
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Triad - Newborn, mother and father: The study involves triads of mother, father, moderately/late preterm born infant, admitted to the NICU. The population of moderately preterm infants admitted to a Neonatal Intensive Care Unit (NICU) and their parents are individuals who face a unique and complex set of challenges. These infants are at a stage when many of their organs and body systems are not yet fully developed. This incomplete development makes them particularly vulnerable to various medical complications.
  As for the parents of these infants, the experience of having a baby admitted to the NICU is often a source of great emotional and psychological stress. Preterm birth, which is generally unexpected, can generate feelings of anxiety, fear and uncertainty about their baby's short- and long-term health. They need clear and understandable informational support to help them feel more involved and less helpless in their baby's care.
  Interventions: Other: Neurobehavioral states and physiological parameters evaluation; Other: Maternal vocal pitch evaluation to assess depressive/anxious state

INTERVENTIONS:
Other: Neurobehavioral states and physiological parameters evaluation — Each individual infant included in the study will be assessed 3 times a week for at least two weeks: specifically, two detections of neurobehavioral states in response to interaction with the mother, two detections with the father, and two detections with the nurse(s) will be made.
  For each infant involved in the study, an audio/video recording of cradle movements and vocalizations will be made at 3 different consecutive times (5 minutes each): baseline; recording during interaction with either parent or nurse; post-interaction assessment.
  The parent or nurse is asked to interact freely with the baby, choosing whether to use voice and touch or only one of the sensory stimulation channels. During the interactions, parents and nurse will in turn be assessed relative to some basic physiological parameters through the use of a band applied to the chest; the infant's physiological parameters during the 3 times will also be recorded.
Other: Maternal vocal pitch evaluation to assess depressive/anxious state — Regarding the assessment of any depressive/anxious states of the mother, as an additional support to the self-report questionnaires the maternal vocal pitch will be specifically assessed through the "Talking about" software (AI algorithm applied to maternal postpartum depression research).

SUMMARY:
The present research project aims to explore the value that contact relationships between caregivers and the preterm infant may have in terms of promoting developmental and maturational processes,by attending to the neurobehavioral states of the infant in response to maternal and paternal voice.

The study is aimed at furthering the still underdeveloped knowledge regarding the possible effects of the paternal voice on the neurobehavioral states of the preterm infant in the crib, comparing them with the effects of exposure to the maternal voice and the voice of a familiar but non-parental figure, such as the NICU nurse.

These behavioral states will also be observed as a function of the psychological condition of the parents, investigating the presence of a possible postpartum depressive condition and/or anxiety of the mother and symptomatology attributable to perinatal affective disorders in the fathers, which are often overlooked; and again, the neurobehavioral responses of the infants will be correlated with the neurophysiological responses of the parents/nurses who interact with them through voice and touch.

The research aims to have a direct impact on both parents and health care personnel: in addition to questionnaires dedicated to screening parents for perinatal psychological disorders, artificial intelligence systems will be used to intercept possible postpartum depression early by recording the maternal voice, enabling the activation of a psychological support intervention and reducing the negative impact that a postpartum depression has on the early mother-child relationship. In addition, information on parent-child interactive modalities will be able to further guide the intake of assignment and particularly the accompaniment of parents during the time of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* For infants: Infants with gestational age between 33 and 36 weeks, weighing around 2kg (LBW - low birth weight), in whom life-threatening conditions have been averted and in stable medical condition will be included in the study.
* For parents: Male and female adults aged between 18 and 50 years.

Exclusion Criteria:

* For infants: Presence of congenital anomalies, neurological disorders, genetic syndromes, and any other condition of developmental atypicality.
* For parents: Parents under 18 years of age; Parents with diagnosed psychiatric disorders and/or sensory disabilities; single parents.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parents and infants born moderately preterm admitted to the NICU experience an unique and complex condition. Babies born moderately preterm, often present challenges related to their not-yet-complete development. The may have organs not yet fully developed resulting in face respiratory and nutritional difficulties. They may have also problems maintaining a stable body temperature, requiring the use of incubators. The high risk of infection is due to their immature immune systems, requiring a sterile and controlled environment. For parents, the long course of intensive care is an extremely stressful and anxiety-provoking experience. Many parents feel overwhelmed by fear and anxiety, and sometimes feel a sense of guilt or responsibility.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal Behavioural Assessment Scale (NBAS) | It takes about 20-30 minutes to administer
  The NBAS is best described as a neurobehavioral assessment scale, designed to describe the newborn's behavioral responses to his/her new extrauterine environment and to document the contribution of the newborn infant to the development of the emerging parent-child relationship. It assesses the newborn's behavioral repertoire with 28 behavioral items, each scored on a 9-point scale. It also includes an assessment of the infant's neurological status on 20 items, each scored on a 4-point scale. It is used to examine the effects of prematurity, low birthweight, undernutrition and a range of pre-and perinatal risk factors, the effects of prenatal substance exposure. The exam does not yield a single score but instead assesses the baby's capabilities across different developmental areas and describes how the baby integrates these areas as s/he deals with her/his new environment.
Edinburgh Postnatal Depression Scale (EPDS) | The tool takes approximately 5 minutes to complete
  The EPDS is the most widely used tool for the screening of perinatal affective disorders during the transition to parenthood. It consists of 10 questions related to various symptoms of depression. The questions on the EPDS focus on depressed mood, anxiety and anhedonia. The EPDS has been constructed to assess depressive symptoms in postpartum women, but it can be used to make extremely fast screening in men who are experiencing the transition to parenthood.
  The response format is a 4-point Likert scale (0 to 3), with an overall score between 0 and 30. A total score of greater than 10 indicates possible depression for mothers, whereas the optimal cutoff for fathers is 12/13.

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Tartarisco, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB)-National Reasearch Council (CNR), Messina 98164, Italy, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egmose I, Vaever MS, Smith-Nielsen J, Varni G, Koppe S. Motor activity and spatial proximity: Relationships to infant emotions and maternal postpartum depression. Infant Behav Dev. 2019 Nov;57:101335. doi: 10.1016/j.infbeh.2019.101335. Epub 2019 Jun 27. PMID 31254811
- [Background] Feldman, R. (2007). Parent-Infant Synchrony: Biological Foundations and Developmental Outcomes. Current Directions in Psychological Science, 16(6), 340-345. doi: 10.1111/j.1467-8721.2007.00532
- [Background] Lee H, White-Traut R. Physiologic responses of preterm infants to the male and female voice in the NICU. J Pediatr Nurs. 2014 Jan-Feb;29(1):e3-5. doi: 10.1016/j.pedn.2013.04.007. Epub 2013 May 14. PMID 23685267
- [Background] Provenzi L, Broso S, Montirosso R. Do mothers sound good? A systematic review of the effects of maternal voice exposure on preterm infants' development. Neurosci Biobehav Rev. 2018 May;88:42-50. doi: 10.1016/j.neubiorev.2018.03.009. Epub 2018 Mar 10. PMID 29535067
- [Background] Saliba S, Gratier M, Filippa M, Devouche E, Esseily R (2020). Fathers' and Mothers' Infant Directed Speech Infuences Preterm Infant Behavioral State in the NICU. Journal of Nonverbal Behavior, 44:437-451. Doi: 10.1007/s10919-020-00335-1